CLINICAL TRIAL: NCT07077135
Title: Transcutaneous Vagal Nerve Stimulation to Treat Disorders of Consciousness
Brief Title: Vagal Nerve Stimulation to Treat Disorders of Consciousness
Acronym: REVELATION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVELATION; NCT06681168 (obsolete NCT alias)
Record Dates: First submitted 2025-05-16; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Disorder of Consciousness
Keywords: vagal nerve stimulation; transcutaneous; auricolar; disorder of consciousness; coma
MeSH Terms: conditions — Consciousness Disorders; Coma | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulated group (Experimental): taVNS stimulation using the Parasym device or sham stimulation will be applied from the time of enrolment (between 7 to 15 days since admission in ICU) until day 90 post-enrolment. Active stimulations will be carried out daily for 60 minutes twice daily during the acute phase and daily during the rehabilitation phase The stimulation waveform includes trains of pulses with widths of 200 µs and repetition rate of 20 Hz (Nurosym proprietary waveform); current delivery will be set at a predefined therapeutic level below 0.25 W/cm² (Watts per centimeter squared), that being the defined risk threshold for a thermal burn. The device adjusts stimulation intensity at 0.8 mA steps; the starting intensity will be set at 16 mA (level 20).
  Interventions: Device: stimulated group
- Control group (Sham Comparator): The Parasym device will be positioned on the patients as for the stimulated group (60 minutes twice daily during the acute phase - two sessions, one in the morning and one in the afternoon), and once daily (single session) during the rehabilitation phase but it won't be switched on.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: stimulated group — Participants will be randomly assigned to receive either taVNS applied to the tragus of the ear or a sham stimulation from the time of randomization for 90 days. Active simulations will be carried out daily using the Parasym device for 60 minutes twice daily during the acute phase (two sessions, one in the morning and one in the afternoon), and once daily (single session) during the rehabilitation phase. The stimulation waveform includes trains of pulses with widths of 200 µs and repetition rate of 20 Hz (Nurosym proprietary waveform); current delivery will be set at a predefined therapeutic level below 0.25 W/cm² (Watts per centimeter squared), that being the defined risk threshold for a thermal burn. The device adjusts stimulation intensity at 0.8 mA steps; the starting intensity will be set at 16 mA (level 20).
  Other Names: experimental arm
  Arms: Stimulated group
Device: Sham (No Treatment) — The sham stimulation involves placing the electrode on the same site without delivering any electrical current. The device will be applied to the tragus without electrical current delivered from the time of randomization for 90 days (i.e., the time of randomization coincides with the first stimulation session).
  Other Names: control group
  Arms: Control group

SUMMARY:
This interventional study aims to assess the clinical efficacy of transcutaneous auricular vagal nerve stimulation (taVNS) against sham stimulation on the recovery of consciousness in patients with disorders of consciousness. The main question it aims to answer is: will taVNS improve patients' behavioral scores or will it produce an improvement in the diagnosed level of consciousness? Researchers will compare the results with non-stimulated unconscious patients to see if the re-gain of consciousness is faster in the treated group.

Participants will undergo taVNS stimulation using the Parasym device or sham stimulation will be applied from the time of enrolment.

Active stimulations will be carried out for 60 minutes twice daily during the acute phase and daily during the rehabilitation phase.

DETAILED DESCRIPTION:
This is a prospective, multicentric, double-blind, parallel, 2 arms, randomized controlled trial that compares active taVNS stimulation against sham stimulation.

The primary objective of this study is to assess the clinical efficacy of transcutaneous auricular vagal nerve stimulation (taVNS) against sham stimulation on the recovery of consciousness in patients with disorders of consciousness (DoC), including comatose patients, unresponsive wakefulness syndrome (UWS) or minimally conscious state (MCS). The hypothesis is that taVNS will improve patients' behavioral scores compared to sham stimulation, as measured by an improvement of at least 3 points in the Coma Recovery Scale-Revised score (CRS-R) or an improvement in the diagnosed level of consciousness, measured at 3 months post-randomization, coinciding with the end of stimulation.

As a secondary objective, we will investigate whether:

1. taVNS is effective in achieving a faster time to recovery of consciousness in DoC patients compared to controls;
2. the CRS-R score differs in the two groups at 3 and 6 months post-randomization;
3. the persistence of improvements in the treated group also at 6 months post-randomization.

taVNS stimulation using the Parasym device or sham stimulation will be applied from the time of enrolment (between 7 to 15 days since admission in ICU) un-til day 90 post-enrolment.

Active stimulations will be carried out daily for 60 minutes twice daily during the acute phase and daily during the rehabilitation phase The stimulation waveform includes trains of pulses with widths of 200 µs and repetition rate of 20 Hz (Nurosym proprietary waveform); current delivery will be set at a prede-fined therapeutic level below 0.25 W/cm² (Watts per centimeter squared), that being the defined risk threshold for a thermal burn. The device adjusts stimulation intensity at 0.8 mA steps; the starting intensity will be set at 16 mA (level 20).

Assuming a delta of response of 30% at 3 months between the experimental and the sham group and considering a 1:1 randomization ratio and a 20% drop-out rate, a sample of 53 patients per group (106 in total) is required to reach a power of 80% (alpha=5% and two-sided test on proportion).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* any acquired cerebral damage of any known etiology;
* diagnosis of coma, UWS, or MCS with the corresponding basal CRS-R (Coma Recovery Scale-Revised) score performed during the screening period from 7 to 15 days since admission in ICU;
* intact ear skin;
* availability of the device.

Exclusion Criteria:

* Patients with severe hemodynamic, respiratory, infectious, or neurological instability requiring active treatment requiring mechanical ventilation or vasoactive drugs or pending acute neurosurgical interventions;
* Need for deep sedation, including general anesthetics (e.g., propofol) or a combination of central-acting sedatives;
* Documented pregnancy;
* Active implant (e.g., pacemaker, cochlear implant);
* History of previous serious neurological disability before the brain injury;
* Seizures or status epilepticus as cause sustaining the disorder of consciousness;
* Patients already enrolled in another ongoing interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of response to stimulation | 90 days post-randomization
  A response is defined as an increase of at least 3 points in the Coma Recovery Scale-Revised (CRS-R), or a clinical change in the diagnosed level of consciousness: from coma to unresponsive wakefulness syndrome (UWS), from UWS to minimally conscious state (MCS), or emergence from MCS. Clinical markers for the diagnostic improvements are derived from the CRS-R scale: • The transition from coma to UWS will be defined as the appearance of eyes opening. • The MCS minus state will be defined by the appearance of visual pursuit, object localization, automatic motor responses, or object manipulation. • The MCS plus will be defined by the appearance of non-functional intentional communication, intelligible verbalization, object recognition, or movement to command. • Emergence from MCS will be defined by the appearance of functional accurate communication or functional object use.

SECONDARY OUTCOMES:
taVNS efficacy in speeding the time of recovery from the disorder of consciousness | 90 days post-randomization
  To evaluate whether taVNS is effective in achieving a faster time to recovery of consciousness in DoC patients compared to controls.
CRS-R score difference | 90 days and 180 days post randomization
  To evaluate if the coma recovery scale revised score (CRS-R) differs in the two groups at 3 and 6 months post-randomization. The CRS-R scale is a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness, and is intended to be used to establish diagnosis, monitor behavioral recovery, predict outcome, and assess treatment effectiveness. It consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level. Minimum score: 0 - Maximum score: 23.
  While the CRS-R total score should not be relied upon to establish a diagnosis, a total score of 10 or greater indicates a diagnosis of MCS or eMCS. The CRS-R can also be used to differentiate patients into "MCS+" and "MCS-" subgroups, based on the presence or absence of receptive or expressive language function.
Efficacy duration | 180 days post-randomization
  To evaluate if improvements persist in the treated group

OTHER OUTCOMES:
Responders phenotype | 180 days
  To evaluate the phenotype of clinical responders by identifying factors after stratification of patients by clinical diagnosis (different etiology, such as traumatic brain injury, subarachnoid hemorrhage, versus intracranial hemorrhage, or ischemic/hemorrhagic stroke).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, MD, Full Professor, Principal Investigator — University of Milano-Bicocca / Fondazione IRCCS San Gerardo dei Tintori; Alberto Addis, MD, Study Director — Fondazione IRCCS San Gerardo dei Tintori
Locations (11):
- Italy (11):
  - ASST degli Spedali Civili di Brescia, Brescia, BS
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - ASST Papa Giovanni XXIII, Bergamo
  - ASST Lariana Ospedale S. Anna, Como
  - Ospedale Policlinico San Martino IRCCS, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Università di Padova, Padua
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Humanitas Research Hospital, Rozzano
  - ASST Sette Laghi Ospedale di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: Yes
Patients recruited in this study cannot provide informed consent at the time of recruitment. The responsible research staff will act as Consultee and consent-eligible patients after discussion with the next-of-kin.
  If the patient has a Power of Attorney or a Legal tutor, he/she will act as a Consultee and will be asked to consent/decline participation in the study on legal behalf of the patient.
  If patients have an Advance Decision Plan, including participation in research studies, the Plan will be respected, and recruitment pursued/abandoned accordingly.
  At follow-up, patients who have regained capacity will be asked to provide Informed Consent and will be given the possibility to:
  * Provide Informed Consent for the acute data and follow-up.
  * Deny research participation and request destruction of acute data collected. Furthermore, participants, their legal representatives, or substitute decision-makers may withdraw consent and discontinue participation at any time during the study.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Result] Sanz LRD, Laureys S, Gosseries O. Towards modern post-coma care based on neuroscientific evidence. Int J Clin Health Psychol. 2023 Jul-Sep;23(3):100370. doi: 10.1016/j.ijchp.2023.100370. Epub 2023 Feb 3. PMID 36817874
- [Result] Vitello MM, Briand MM, Ledoux D, Annen J, El Tahry R, Laureys S, Martin D, Gosseries O, Thibaut A. Transcutaneous vagal nerve stimulation to treat disorders of consciousness: Protocol for a double-blind randomized controlled trial. Int J Clin Health Psychol. 2023 Apr-Jun;23(2):100360. doi: 10.1016/j.ijchp.2022.100360. Epub 2022 Nov 29. PMID 36467262
- [Result] Urbin MA, Lafe CW, Simpson TW, Wittenberg GF, Chandrasekaran B, Weber DJ. Electrical stimulation of the external ear acutely activates noradrenergic mechanisms in humans. Brain Stimul. 2021 Jul-Aug;14(4):990-1001. doi: 10.1016/j.brs.2021.06.002. Epub 2021 Jun 18. PMID 34154980
- [Result] Briand MM, Gosseries O, Staumont B, Laureys S, Thibaut A. Transcutaneous Auricular Vagal Nerve Stimulation and Disorders of Consciousness: A Hypothesis for Mechanisms of Action. Front Neurol. 2020 Aug 25;11:933. doi: 10.3389/fneur.2020.00933. eCollection 2020. PMID 32982941
- [Result] Sharon O, Fahoum F, Nir Y. Transcutaneous Vagus Nerve Stimulation in Humans Induces Pupil Dilation and Attenuates Alpha Oscillations. J Neurosci. 2021 Jan 13;41(2):320-330. doi: 10.1523/JNEUROSCI.1361-20.2020. Epub 2020 Nov 19. PMID 33214317
- [Result] Gerges ANH, Williams EER, Hillier S, Uy J, Hamilton T, Chamberlain S, Hordacre B. Clinical application of transcutaneous auricular vagus nerve stimulation: a scoping review. Disabil Rehabil. 2024 Dec;46(24):5730-5760. doi: 10.1080/09638288.2024.2313123. Epub 2024 Feb 16. PMID 38362860
- [Result] Wu X, Xie L, Lei J, Yao J, Li J, Ruan L, Hong J, Zheng G, Cheng Y, Long L, Wang J, Huang C, Xie Q, Zhang X, He J, Yu X, Lv S, Sun Z, Liu D, Li X, Zhu J, Yang X, Wang D, Bao Y, Maas AIR, Menon D, Xue Y, Jiang J, Feng J, Gao G; ACES Participants. Acute traumatic coma awakening by right median nerve electrical stimulation: a randomised controlled trial. Intensive Care Med. 2023 Jun;49(6):633-644. doi: 10.1007/s00134-023-07072-1. Epub 2023 May 13. PMID 37178149
- [Result] Schiff ND. Recovery of consciousness after brain injury: a mesocircuit hypothesis. Trends Neurosci. 2010 Jan;33(1):1-9. doi: 10.1016/j.tins.2009.11.002. Epub 2009 Dec 1. PMID 19954851
- [Result] Manta S, Dong J, Debonnel G, Blier P. Optimization of vagus nerve stimulation parameters using the firing activity of serotonin neurons in the rat dorsal raphe. Eur Neuropsychopharmacol. 2009 Apr;19(4):250-5. doi: 10.1016/j.euroneuro.2008.12.001. Epub 2009 Jan 15. PMID 19150228
- [Result] Sandroni C, Citerio G, Taccone FS. Automated pupillometry in intensive care. Intensive Care Med. 2022 Oct;48(10):1467-1470. doi: 10.1007/s00134-022-06772-4. Epub 2022 Jun 30. No abstract available. PMID 35773500
- [Result] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Practice Guideline Update Recommendations Summary: Disorders of Consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Arch Phys Med Rehabil. 2018 Sep;99(9):1699-1709. doi: 10.1016/j.apmr.2018.07.001. Epub 2018 Aug 8. PMID 30098791